CLINICAL TRIAL: NCT04818203
Title: A Single Center, Randomized, Evaluator and Subject Blind, Placebo Controlled, Parallel, Phase 1/2 Study for the Anti-wrinkle Efficacy Assessment and Safety Evaluation by Treating Cluster of Autologous Dermal Fibroblasts, 3D-F in Patients With Bilateral Crow's Feet
Brief Title: A Study on the Anti-Wrinkle Efficacy Assessment and Safety Evaluation of the Cluster of Autologous Dermal Fibroblast on Bilateral Crow's Feet
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: S.Biomedics Co., Ltd. (Industry)
Collaborators: Dt&Sanomedics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SB-FC-001
Record Dates: First submitted 2021-03-23; First posted 2021-03-26 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Crow's Feet
Keywords: Fibroblast; Anti-Wrinkle; Cell therapy; Cell spheroid; S.Biomedics

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test Group (Experimental): Participants receive 1 mL of clusters of autologous dermal fibroblast to three spots around the left eye and three spots around the right eye along the periorbital wrinkles on both sides, perpendicularly to the wrinkles.
  Interventions: Biological: Clusters of Autologous Dermal Fibroblasts
- Placebo (Placebo Comparator): Participants receive 1 mL of placebo solution to three spots around the left eye and three spots around the right eye along the periorbital wrinkles on both sides, perpendicularly to the wrinkles.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Clusters of Autologous Dermal Fibroblasts — Dose: 1 x 10^7 cells/1 mL/vial
  Other Names: 3D-F; FECS-DF
  Arms: Test Group
Other: Placebo — The injection solution without clusters of autologous dermal fibroblasts
  Arms: Placebo

SUMMARY:
This study is a phase 1/2 clinical trial to evaluate the safety and efficacy of administering clusters of autologous dermal fibroblasts to subjects with periorbital wrinkles on both sides.

If subjects who have signed the Informed consent form voluntarily are enrolled in this study, they will be tested for eligibility during the screening period. Subjects will visit the study site a total of 6 times while participating in this study. The subjects who meet the inclusion/exclusion criteria will receive a total of one dose of the IP (Visit 3). Then, the efficacy evaluation will be conducted at Visit 4 (Week 2), Visit 5 (Week 12), and Visit 6 (Week 24), and safety will also be evaluated at each visit.

DETAILED DESCRIPTION:
This study is a phase 1/2 clinical trial in patients with periorbital wrinkles on both sides. The study consists of phase 1 to evaluate safety and phase 2 to evaluate efficacy.

* Phase 1: Single center, randomized, placebo-controlled, parallel design. If a subject voluntarily signs the written informed consent form to participate in this study, he/she will be enrolled as a subject after eligibility evaluation. After a single administration of the study drug to a subject, safety and efficacy will be evaluated at Week 2, Week 12, and Week 24 visits after administration.

If an adverse drug reaction of grade 3 or higher occurs in 3 subjects 2 weeks after administration of the study drug in the phase 1 study; if an adverse drug reaction occurs in 0/3 subjects, the phase 2 study will be conducted after completing the phase 1 study; if an adverse drug reaction occurs in 2/3 or more subjects, the study will be terminated; and if an adverse drug reaction occurs in 1/3 subjects, 3 additional subjects will be enrolled to proceed with the study. After the safety of subjects in the phase 1 study is confirmed by Week 12, the phase 2 study will be conducted.

* Phase 2: Single center, randomized, subject- and assessor- blinded, placebo controlled, parallel design.

If safety is secured 12 weeks after administering the study drug in phase 1, phase 2 will be conducted.

Only the subjects that meet the final inclusion criteria will be assigned sequentially and recognized by the same procedure and will receive the study drug once.

Safety and efficacy will be evaluated at Week 2, Week 12, Week 24 after administration. All subjects will be tested on the same schedule.

ELIGIBILITY:
Inclusion Criteria:

* Participants of ages 19 and older
* Those with at least 3 points (Moderate) of the IGA-LCL severity scale on both sides in the rest state during screening
* Those who have visually symmetrical periorbital wrinkles on both sides and have the same IGA-LCL severity scale score in the rest state
* Those who agreed to discontinue all dermatological treatments including facial wrinkle improvement during this study period
* Subjects with healthy and undamaged skin at the sampling area (e.g., behind the ears, inside of the arms, armpits, groin, etc.)
* Those who meet the following criteria based on the blood test at screening or baseline visits

  * White Blood Cell : ≥4.5x10^3/μl and ≤11.0x10^3/μl
  * Platelet count : ≥100x10^3/μl
  * Hemoglobin : ≥9 g/dL
* Those who sign the written consent form after hearing the explanation of the purpose, method, and efficacy of this study
* Those who can be followed up during the study period

Exclusion Criteria:

* Those with arterial bleeding or severe variceal bleeding in the body
* Those with hypersensitivity to bovine protein or gentamicin
* Pregnant and breast-feeding or who planning to conceive within six months of clinical trial medication
* Out of who are pregnant or breast-feeding and A woman who is likely to be pregnant in a postmenopausal or a state of non-Infertility surgery and men with reproductive abilities not willing or planning to use the appropriate contraception defined in this clinical trial during their participation in clinical trials
* Those with or suspected of having autoimmune diseases (e.g., myasthenia gravis, systemic lupus erythematosus, rheumatoid arthritis, etc.)
* At the screening visit, patients with chronic skin disease or such a medical history
* Those with a medical history or a positive test result for any of the following: hepatitis C virus antibody (HCV Ab), hepatitis B surface antigen (HBsAg), human immunodeficiency virus-1 (HIV-1) antibody, human immunodeficiency virus-2 (HIV-2) antibody (However, if HCV is proven to be completely cured based on the HCV RNA test, he/she can be enrolled as a subject.)
* Those with severe heart diseases (e.g., myocardial infarction, heart failure, etc.) or severe liver diseases (e.g., hepatocirrhosis, liver failure, etc.) or severe kidney diseases (e.g., renal failure, etc.)
* Those who have tumors or have such medical history within 5 years of screening (However, if the malignant tumor does not relapse for more than 5 years, the candidate may be enrolled as a subject, and in the case of basal cell carcinoma or intradermal squamous cell carcinoma that does not relapse after resection, he/she can be enrolled as a subject.)
* Those with genetic diseases affecting fibroblast or collagen
* Those who have undergone anticoagulant therapy or antiplatelet therapy within 10 days prior to administration of the study drug, or those who are expected to need to receive them within 3 days after administration of the study drug (However, if the drug is being administered at the time of screening, it is possible to participate in the clinical trial after a seven-day not administering medication period only if the temporary suspension does not pose a medical risk under the tester's judgment, tried tissue biopsy Schedule.)
* Those who have active or infectious skin diseases (skin infection, inflammation, herpes, etc.), keloids, unhealed wounds or scars, tumors, etc. at the site where the study drug will be administered, or those who have previously received radiation treatment
* Those with hypersensitivity to local anesthetics (however, those who agree to receive the procedure without applying an anesthetic agent due to hypersensitivity to local anesthetics, do not fall under this criteria.)
* A person who has a history of significant adverse or hypersensitive reactions to the composition of medications for clinical trials
* Those who have undergone procedures that can affect periorbital wrinkles, such as dermabrasion, skin regeneration, and plastic surgery, etc, among facial procedures including the eye area* or those who are expected to have such procedures during the study period
* Those who participated in another study and received an investigational drug or used an investigational medical device within 6 months prior to participation in this study, or those who are scheduled to participate in another study during this study period
* Those with a medical history of autologous dermal fibroblast treatment
* Those with a medical history of anaphylaxis or severe complex allergies
* Those with a medical history of keloid formation, hyperpigmentation, or hypertrophic scars on the face
* Those who have clinically serious disorders in the cardiovascular system, digestive system, respiratory system, endocrine system, or central nervous system, or have had or currently have a mental disorder that significantly affects this study
* Those who received systemic corticosteroid within 12 weeks prior to participation in this study
* Those who refuse to take pictures of the site where the study drug is administered
* Those who are judged to be ineligible by the investigator to participate in this study for other reasons

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2025-07-05 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Improvement rate of 2 points or more of IGA-LCL Wrinkle Severity | Baseline, Week 24
  After independent assessment of IGA-LCL (Investigator's Global Assessment of Lateral Canthal Lines) Wrinkle Severity of the subject's left/right crow's feet in the rest state assessed through photographs, the percentage of subjects who improved by 2 points or more on both sides compared to the baseline are presented by group

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Seoul, South Korea